CLINICAL TRIAL: NCT03339258
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Doxazosin for Nightmares, Sleep Disturbance, and Non-Nightmare Clinical Symptoms in Post-Traumatic Stress
Brief Title: A Randomized Controlled Trial of Doxazosin for Nightmares, Sleep Disturbance, and Non-Nightmare Clinical Symptoms in PTSD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Northern California Institute of Research and Education (Other)
Responsible Party: Principal Investigator, Anne Richards, Staff Psychiatrist, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-17-1-0234
Record Dates: First submitted 2017-11-06; First posted 2017-11-13 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Posttraumatic Stress Disorder; Post-traumatic Stress Disorder; PTSD; Doxazosin; Nightmares; Sleep Disturbance
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias | interventions — Doxazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxazosin Mesylate, Extended Release (Experimental): Subjects will undergo a 4-week titration phase during which doxazosin may be increased to a maximum dose of 10mg at bedtime based on symptoms and tolerability. After the 4-week titration phase, subjects will continue at stable dose of study medication for a 4-week stable dose phase.
  Interventions: Drug: Doxazosin Mesylate, Extended Release
- Placebo (Placebo Comparator): Subjects will undergo a 4-week titration phase during which the placebo may be increased to a maximum dose of 10mg at bedtime based on symptoms and tolerability. After the 4-week titration phase, subjects will continue at stable dose of study placebo for a 4-week stable dose phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin Mesylate, Extended Release — Doxazosin is FDA-approved for the treatment of hypertension and urinary outflow problems associated with benign prostatic hyperplasia. The immediate-release formulation is approved for use from 1mg up to 16mg. Based on drug company information and Micromedex, the SFVA pharmacy on-line reference resource for drug information, the only contraindication to use of doxazosin is hypersensitivity to doxazosin, its contents, or other quinazolines (e.g. prazosin, terazosin).
  Other Names: Cardura XL
  Arms: Doxazosin Mesylate, Extended Release
Drug: Placebo — Placebo, or inactive pill.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled trial of doxazosin will assess doxazosin's effectiveness for PTSD nightmares, subjective sleep quality, and non-nightmare PTSD symptoms in adult men and women veterans with full and partial-syndromal PTSD.

DETAILED DESCRIPTION:
This study will involve a randomized, double-blind, placebo-controlled, flexible dose trial of doxazosin (1-10mg) for PTSD nightmares, sleep disturbance and overall PTSD symptoms. The target sample will consist of 60 male and female subjects with chronic PTSD symptoms and prominent nightmares randomly assigned to receive doxazosin (n=30) or placebo (n=30). Participants will be enrolled at the San Francisco VA Medical Center. Following baseline consent procedures, eligibility assessments, and 1-week of baseline assessments including self-report surveys, actigraphy, and at-home EEG (Sleep Profiler), all subjects will initiate doxazosin or equivalently marked placebo at 1mg at bedtime. Subjects will undergo a 4-week titration phase during which doxazosin or placebo may be increased to a maximum dose of 10mg (or equivalently marked placebo) at bedtime based on symptoms and tolerability. After the 4-week titration phase, subjects will continue at stable dose of study medication for a 4-week stable dose phase. Subjects will be asked to complete sleep diaries daily during their participation in the study. In the last week of the stable dose phase, participants will undergo an additional week of at-home sleep monitoring using actigraphy, complete end of treatment surveys, and undergo end-of-treatment clinical assessments and discontinuation of study medication. After discontinuation of study medication, participants will complete three additional days of sleep diaries.

ELIGIBILITY:
Inclusion Criteria:

* U.S. military veteran or civilian;
* age 18-75 and
* current full syndromal PTS as indexed by the CAPS-5 (Clinician-administered PTSD scale) or have a current CAPS-5 score ≥ 20, and CAPS-IV recurrent distressing dreams item of ≥ 3; or a CAPS-5 score ≥ 12, and CAPS-IV recurrent distressing dream item of ≥ 4.

Exclusion Criteria:

* DSM-5 current moderate to severe alcohol or drug use disorder in the last 3 months; moderate alcohol or drug use disorder in the last 3 months will be reviewed on a case-by-case basis;
* history of any psychiatric disorder with active psychosis or mania in the past 5 years;
* exposure to trauma within the last 3 months;
* prominent suicidal or homicidal ideation;
* score of 16 or greater AHI based on ApneaLink data analysis in the absence of effective sleep treatment (such as CPAP or oral device)
* neurologic disorder or systemic illness affecting central nervous system function;
* chronic or unstable medical illness including unstable angina, myocardial infarction within the past 6 months, congestive heart failure, preexisting hypotension or standing systolic blood pressure < 100 mmHg at eligibility (V0); orthostatic hypotension defined as orthostatic systolic decrease after 3 minutes standing >20 mmHg or any BP decrease accompanied by lightheadedness; complete heart block or arrhythmia on ECG; chronic renal or hepatic failure, and pancreatitis;
* history of priapism or refusal to hold off on as needed phosphodiesterase inhibitors;
* pregnancy, breastfeeding and/or refusal to use effective birth control (female participants);
* previous adverse reaction to an alpha-1-antagonist;
* current use of a medication with alpha-1 blocking properties for insomnia, alpha-1 antagonists, alpha-2 agonists, boceprevir; midodrine; and
* use of yohimbine, Ma huang or other non-FDA approved substances or herbal remedies that the investigators consider pose a risk to participation
* homelessness (includes living in a temporary shelter);
* subjects who, in the opinion of the investigator, are otherwise unsuitable for a study of this type.

Participants taking SSRIs, duloxetine, bupropion, mirtazapine, and venlafaxine may be included if they have been on a stable dose for 4 weeks. Participants may be included if they are in psychotherapy treatment as long as they do not participate in evidence-based trauma-focused or nightmare-focused psychotherapy (such as cognitive processing therapy, prolonged exposure therapy, or imagery rehearsal therapy) while in the trial. Participants who are normotensive and do not have orthostatic hypotension while on stable-dose beta-blocker may be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale (CAPS) Distressing Dream Score | Baseline and Week 9 (end-of-treatment)
  For the assessment of nightmares, the CAPS developed for the DSM-IV will be utilized. The CAPS IV's wide use as an outcome measure in clinical research has provided abundant information about its reliability and responsiveness to change with treatment in general and for nightmares specifically. All existing studies of alpha-blockers for PTS nightmares and non-nightmare symptoms have used the CAPS for DSM-IV, and therefore our results will be more comparable to existing studies. The distressing dreams item from the CAPS for DSM-IV also has strong behavioral anchors, providing detail on both the frequency and intensity of nightmares. A CAPS (DSM-IV) distressing dreams item score of >=3, as used in prior research on alpha-blockers, will be a requirement for inclusion. Change in CAPS distressing dream score between baseline and end-of-treatment will be the primary measure of the reduction of nightmare frequency/intensity.
Change in Pittsburgh Sleep Quality Index (PSQI) | Weeks 0, 1, 3, 6, 9 (end-of-treatment)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Clinical and clinimetric properties of the PSQI were assessed over an 18-month period and acceptable measures of internal homogeneity, consistency (testretest reliability), and validity were obtained. A global PSQI score > 5 yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p 0.001) in distinguishing good and poor sleepers. The clinimetric and clinical properties of the PSQI suggest its utility both in psychiatric clinical practice and research activities.
Change in CAPS PTS Symptom Score | Baseline and Week 9 (end-of-treatment)
  Change in total CAPS score, minus the distressing dreams item score

SECONDARY OUTCOMES:
Change in minutes of wake after sleep onset (WASO) | Daily, weeks 0-8
  Each morning the subject will record the clock times of their sleep onset and offset, number of nighttime awakenings, wake time in minutes after sleep onset (WASO), number of nightmares and intensity of the worst nightmare on a 10-point scale. They will also rate their sleep quality on a scale from 1-100. From this data, measures of TST, WASO, and SM can be calculated.
Change in total sleep time (TST) | Daily, weeks 0-8
  Each morning the subject will record the clock times of their sleep onset and offset, number of nighttime awakenings, wake time in minutes after sleep onset (WASO), number of nightmares and intensity of the worst nightmare on a 10-point scale. They will also rate their sleep quality on a scale from 1-100. From this data, measures of TST, WASO, and SM can be calculated.
Change in sleep maintenance (SM) | Daily, weeks 0-8
  Each morning the subject will record the clock times of their sleep onset and offset, number of nighttime awakenings, wake time in minutes after sleep onset (WASO), number of nightmares and intensity of the worst nightmare on a 10-point scale. They will also rate their sleep quality on a scale from 1-100. From this data, measures of TST, WASO, and SM can be calculated.
Nightmare Distress Questionnaire (NDQ) | Weeks 0, 1, 3, 6, 9 (end-of-treatment)
  The NDQ is a self-report assessment of the degree of distress that nightmares cause, and is shown to be a valid, reliable measure of the effects of nightmares.
PTSD Checklist for DSM- 5 (PCL-5) | Weeks 0, 1, 3, 6, 9 (end-of-treatment)
  The PCL-5 will be used as a secondary measure and to assess the internal consistency of the CAPS PTSD symptom score. The PCL-5 is a validated self-report rating scale for assessing PTSD symptoms. It consists of 20 items that correspond to the DSM-5 symptoms of PTSD.
Objective measure of change in TST | All subjects will wear the actigraph daily for 7 days at pre-treatment baseline (week 0), 7 days in week 5 of study drug treatment, and at end-of-treatment week 8 prior to drug discontinuation.
  The AMI Octagonal Basic Motionlogger (www.ambulatorymonitoring.com), which is worn on the wrist like a watch, is an advanced actigraph which has sufficient memory to record movements for up to 28 days. As indicated by the American Academy of Sleep Medicine Standards of Practice Committee, actigraphy can improve the reliability of self-report estimates of sleep wake timing and may play an important 15 role in the diagnosis and treatment of insomnia. It is also appropriate for the assessment of stability of treatment effects, including the assessment of changes in night-to-night variability in various sleep measures. Our lab has used this actigraph extensively, providing support for its usability in research subjects. High resolution data can be down-sampled for actigraphic sleep-wake estimation.
Objective measure of change in WASO | All subjects will wear the actigraph daily for 7 days at pre-treatment baseline (week 0), 7 days in week 5 of study drug treatment, and at end-of-treatment week 8 prior to drug discontinuation.
  The AMI Octagonal Basic Motionlogger (www.ambulatorymonitoring.com), which is worn on the wrist like a watch, is an advanced actigraph which has sufficient memory to record movements for up to 28 days. As indicated by the American Academy of Sleep Medicine Standards of Practice Committee, actigraphy can improve the reliability of self-report estimates of sleep wake timing and may play an important 15 role in the diagnosis and treatment of insomnia. It is also appropriate for the assessment of stability of treatment effects, including the assessment of changes in night-to-night variability in various sleep measures. Our lab has used this actigraph extensively, providing support for its usability in research subjects. High resolution data can be down-sampled for actigraphic sleep-wake estimation.
Objective measures of change in SM | All subjects will wear the actigraph daily for 7 days at pre-treatment baseline (week 0), 7 days in week 5 of study drug treatment, and at end-of-treatment week 8 prior to drug discontinuation.
  The AMI Octagonal Basic Motionlogger (www.ambulatorymonitoring.com), which is worn on the wrist like a watch, is an advanced actigraph which has sufficient memory to record movements for up to 28 days. As indicated by the American Academy of Sleep Medicine Standards of Practice Committee, actigraphy can improve the reliability of self-report estimates of sleep wake timing and may play an important 15 role in the diagnosis and treatment of insomnia. It is also appropriate for the assessment of stability of treatment effects, including the assessment of changes in night-to-night variability in various sleep measures. Our lab has used this actigraph extensively, providing support for its usability in research subjects. High resolution data can be down-sampled for actigraphic sleep-wake estimation.

OTHER OUTCOMES:
Beck Depression Inventory (BDI) | Weeks 0, 1, 3, 6, and 9 (end-of-treatment)
  The BDI is a widely used self-report measure which includes subjective ratings of 21 depressive symptoms.
Sexual Health Inventory for Men (SHIM) | Weeks 0, 1, 3, 6, and 9 (end-of-treatment)
  The SHIM is a well-validated measure used in urology research, will be utilized to assess the effects of doxazosin on erectile function in men, the aspect of sexual functioning that may be most affected by doxazosin.
Male Sexual Health Questionnaire (MSHQ) | Weeks 0, 1, 3, 6, and 9 (end-of-treatment)
  The MSHQ will be utilized as a more global measure of sexual health, encompassing erectile function, ejaculatory function, and satisfaction in men.
Female Sexual Functioning Index (FSFI) | Weeks 0, 1, 3, 6, and 9 (end-of-treatment)
  The FSFI will be used to assess for various elements of sexual functioning in women, including arousal and satisfaction.
World Health Organization Quality of Life inventory (WHOQOL-BREF) | Weeks 0, 1, 3, 6, and 9 (end-of-treatment)
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument and more convenient for use in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Richards, MD, MPH, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] De Jong J, Wauben P, Huijbrechts I, Oolders H, Haffmans J. Doxazosin treatment for posttraumatic stress disorder. J Clin Psychopharmacol. 2010 Feb;30(1):84-5. doi: 10.1097/JCP.0b013e3181c827ae. No abstract available. PMID 20075659
- [Derived] Richards A, Santistevan AC, Yack LM, West AC, Berg E, Pracar S, Batki SL, Seal KH, Neylan TC. A double-blind, randomized, placebo-controlled trial of doxazosin for posttraumatic distressing dreams and sleep disturbance in men and women with posttraumatic stress. J Clin Sleep Med. 2025 Dec 1;21(12):2165-2179. doi: 10.5664/jcsm.11908. PMID 41042258